CLINICAL TRIAL: NCT07170579
Title: Effects of High-Intensity Interval Training on Functional Fit-ness in Older Adults: A Randomized Controlled
Brief Title: Effects of HIIT in Older Adults
Acronym: HIIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Politécnico de Bragança (Other)
Responsible Party: Principal Investigator, André Schneider, Principal Investigator, Instituto Politécnico de Bragança
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2067313
Record Dates: First submitted 2025-08-28; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Aging
Keywords: High-intensity interval training; functional fitness; older adults; aging; physical exercise; autonomy; activities of daily living
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HIIT Group (Experimental): Participants perform high-intensity interval training (HIIT) sessions three times per week, including aerobic exercises with intervals of effort and recovery, adapted to older adults.
  Interventions: Other: Exercise
- Control Group (No Intervention): Participants maintain their usual daily activities and do not receive any structured exercise intervention during the study period.

INTERVENTIONS:
Other: Exercise — Participants engaged in High-Intensity Interval Training (HIIT) sessions three times per week, each lasting 60 minutes. Sessions included a 10-minute warm-up, a central HIIT block with cycles of aerobic exercises performed at high intensity (30-60 seconds) alternated with active recovery (60-90 seconds), followed by a 10-minute aerobic functional segment and a 10-minute cool-down with stretching. Exercises included modified jumping jacks, stationary marching, high knees, squats, and functional movements tailored to the participants' physical capacity. Training intensity was monitored using the Borg Rating of Perceived Exertion scale, targeting 13-17 during effort phases and 9-11 during recovery.
  Arms: HIIT Group

SUMMARY:
This study investigated the effects of high-intensity interval training (HIIT) on functional fitness in older adults. As people age, they often experience a natural decline in physical abilities such as strength, flexibility, balance, and endurance, which can limit their ability to perform daily activities independently. Finding safe and effective exercise strategies to maintain or improve these abilities is critical for promoting healthy aging and preserving autonomy.

In this study, older adults participated in a structured HIIT program adapted to their functional capacity. HIIT consists of short bursts of intense physical activity followed by periods of active rest. This type of training is known for improving cardiovascular and muscular fitness in a short period of time.

Participants were assessed on various aspects of physical function before, during, and after the intervention. Tests included handgrip strength, upper and lower body strength, flexibility, aerobic endurance, and mobility.

The results showed that HIIT significantly improved physical function in older adults, including increased muscle strength, flexibility, aerobic capacity, and agility. These findings suggest that HIIT can be a safe, efficient, and accessible option to promote health and independence in the aging population.

DETAILED DESCRIPTION:
This randomized controlled study aimed to evaluate the effectiveness of a high-intensity interval training (HIIT) protocol on functional fitness in community-dwelling older adults. With the global rise in life expectancy and the associated functional decline in aging populations, there is an increasing demand for time-efficient, evidence-based interventions that can promote physical independence and healthy aging.

Participants aged 60 years or older were recruited and assigned to either a HIIT intervention group or a control group. The HIIT group engaged in supervised training sessions three times per week. Each session included a warm-up, a core HIIT segment with short bursts of high-intensity movements interspersed with active recovery, followed by a cool-down. Exercises were adapted to be safe and appropriate for older adults, focusing on full-body functional movements and performed in a group setting under professional supervision.

Functional fitness was evaluated using the Senior Fitness Test battery and handgrip strength testing. This included assessments of:

* Lower body strength (30-second chair stand)
* Upper body strength (arm curl test)
* Lower body flexibility (chair sit-and-reach)
* Upper body flexibility (back scratch test)
* Agility and dynamic balance (Timed Up and Go test)
* Cardiorespiratory endurance (2-minute step test)
* Handgrip strength (digital dynamometer, dominant hand)

Measurements were taken at three time points: pre-intervention (M1), midpoint (M2), and post-intervention (M3). Statistical analysis included nonparametric ANOVA-type models (Brunner-Langer), given the non-normal distribution of many outcome variables.

The results indicated statistically significant improvements in the HIIT group for several domains of functional fitness compared to the control group. Notably, participants in the HIIT group showed:

* Increased handgrip strength
* Improved upper and lower limb flexibility
* Enhanced aerobic endurance
* Improved mobility and agility (TUG test)
* Increased upper body strength (arm curl)

These results support the effectiveness of HIIT in improving multiple aspects of physical function among older adults, without the need for resistance machines or prolonged exercise sessions. The findings highlight the feasibility and clinical relevance of using HIIT as a tool to enhance physical independence, prevent disability, and reduce the burden on health systems.

All procedures were approved by the Ethics Committee of the Polytechnic Institute of Bragança and followed international guidelines (SPIRIT, CONSORT, Declaration of Helsinki). Participation was voluntary, and informed consent was obtained from all individuals.

ELIGIBILITY:
Inclusion Criteria:

* Community-dwelling individuals aged 60 years or older
* Able to walk independently without assistive devices
* Sufficient cognitive ability to follow instructions and participate in assessments
* Medically stable and cleared for physical activity by a healthcare provider
* No current participation in structured exercise programs
* Willingness to participate in the intervention and attend scheduled assessments
* Provided written informed consent

Exclusion Criteria:

* Individuals younger than 60 years
* Severe musculoskeletal, cardiovascular, or neurological conditions that contraindicate physical exercise
* Uncontrolled hypertension or diabetes
* Recent surgery or hospitalization in the past 6 months
* Severe visual or auditory impairments that limit test performance
* Use of mobility aids (e.g., walker or cane for ambulation)
* Participation in another clinical trial simultaneously

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-08-20 (Actual)

PRIMARY OUTCOMES:
Number of steps completed in the 2-Minute Step Test | Baseline (Week 0), Mid-intervention (Week 33), and Post-intervention (Week 65)
  Number of steps completed in the 2-Minute Step Test The 2-Minute Step Test assesses aerobic endurance. Participants are instructed to march in place for two minutes, raising the knees to a target height midway between the kneecap and hip. The number of steps completed with the right knee reaching the target is counted.

SECONDARY OUTCOMES:
Handgrip strength (kg) | Baseline (Week 0), Mid-intervention (Week 33), and Post-intervention (Week 65)
  Maximal isometric strength of the dominant hand measured using a digital handgrip dynamometer (JAMAR®). Participants performed three attempts with 30-second rest intervals; the highest value was recorded.
Upper body strength (Arm Curl Test) | Baseline (Week 0), Mid-intervention (Week 33), and Post-intervention (Week 65)
  Number of repetitions performed using a 2 kg dumbbell (women) or 3 kg (men) in 30 seconds, with the dominant arm.
Lower body strength (30-Second Chair Stand) | Baseline (Week 0), Mid-intervention (Week 33), and Post-intervention (Week 65)
  Number of full sit-to-stand repetitions completed in 30 seconds, without using arms.
Upper body flexibility (Back Scratch Test) | Baseline (Week 0), Mid-intervention (Week 33), and Post-intervention (Week 65)
  Distance (in cm) between the middle fingers when reaching behind the back, one hand over the shoulder and the other up the middle of the back.
Lower body flexibility (Chair Sit-and-Reach Test) | Baseline (Week 0), Mid-intervention (Week 33), and Post-intervention (Week 65)
  Distance (in cm) from fingertips to toes while sitting on a chair and reaching toward the foot with one leg extended.
Agility and dynamic balance (Timed Up and Go Test - TUG) | Baseline (Week 0), Mid-intervention (Week 33), and Post-intervention (Week 65)
  Time (in seconds) taken to rise from a chair, walk 3 meters, turn, return, and sit down again.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Politécnico de Bragança, Bragança, Portugal

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/79/NCT07170579/ICF_000.pdf